CLINICAL TRIAL: NCT00371410
Title: The Safety and the Efficacy of Combined Vitrectomy, Intravitreal Triamcinolone Acetonide and Macular Focal Laser Photocoagulation for the Treatment of Intractable Diffuse Diabetic Macular Edema
Brief Title: Sequentially Combined Vitrectomy, IVTA and Macular Focal Laser Photocoagulation for Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-05-029
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-08

CONDITIONS: Diabetic Macular Edema
Keywords: Vitrectomy; Intravitreal triamcinolone acetonide; Macular focal laser photocoagulation; Best-corrected visual acuity; Central macular thickness
MeSH Terms: interventions — Vitrectomy

INTERVENTIONS:
Procedure: vitrectomy
Drug: intravitreal triamcinolone acetonide
Procedure: macular focal laser photocoagulation

SUMMARY:
Macular edema constitutes the primary cause of visual impairment in diabetic patients with a disease duration of 20 years or more. Intravitreal triamcinolone (IVTA) and macular focal laser photocoagulation were reported to generate favorable results in the treatment of diabetic macular edema, but there have been patients with diffuse diabetic macular edema refractory to such treatment modalities. The present study will test the safety and the efficacy of the combined treatment of vitrectomy, IVTA and macular focal laser photocoagulation in the treatment of intractable diffuse diabetic macular edema.

DETAILED DESCRIPTION:
Fifty eyes from 50 diabetic patients were included, who had been diagnosed with intractable diffuse diabetic macular edema (DME). Intractable diffuse DME was defined as a biomicroscopically, angiographically and tomographically proven diffuse DME, which did not respond to or recurred after the previous intravitreal triamcinolone acetonide (IVTA) and/or macular focal laser photocoagulation. The central macular thickness (CMT) had to be greater than 250 μm. Preoperative ocular examination included best corrected visual acuity (BCVA) using the ETDRS chart, applanation tonometry, slit-lamp biomicroscopy, dilated fundus examination, optical coherence tomography (OCT) and fluorescein angiography. Pars plana vitrectomy with removal of retinal internal limiting membrane (ILM) was performed in all the 50 subject eyes. On the day after vitrectomy, triamcinolone acetonide (0.1 mL, 40 mg/mL) was injected intravitreally. Macular focal laser photocoagulation was performed 2 weeks after vitrectomy. As main outcome measures, BCVA was recorded and the CMT was measured using OCT by independent observers for all subjects at 3 and 6 months after the laser photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes mellitus
* intractable diffuse DME (diffuse DME which did not respond to or recurred after the previous IVTA and/or macular focal laser photocoagulation)
* the central macular thickness (CMT) greater than 250 μm

Exclusion Criteria:

* presence of vitreomacular traction
* a prior history of treatment for the DME within 3 months or vitreoretinal surgery

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2007-10

PRIMARY OUTCOMES:
Best-corrected visual acuity
Central macular thickness

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, MD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kang SW, Park SC, Cho HY, Kang JH. Triple therapy of vitrectomy, intravitreal triamcinolone, and macular laser photocoagulation for intractable diabetic macular edema. Am J Ophthalmol. 2007 Dec;144(6):878-885. doi: 10.1016/j.ajo.2007.07.044. Epub 2007 Oct 15. PMID 17936715